CLINICAL TRIAL: NCT01381770
Title: Platelet-derived Factors for Treatment of Muscular Lesions: a Phase II Trial
Brief Title: Platelet-derived Factors for Treatment of Muscular Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Claudio Pavesi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: plt-msl001
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Muscle Lesions
Keywords: muscular lesions grade 2; muscular lesions grade 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platelet-derived repairing factors (Experimental)
  Interventions: Biological: platelet-derived repairing factors

INTERVENTIONS:
Biological: platelet-derived repairing factors — autologous platelet lysate injection within 24 hours from lesion

SUMMARY:
The purpose of this study is to demonstrate that platelet-derived repairing factors are effective and safe in the treatment of muscular lesion grade 2 or 3, a Phase II, open-label, single arm, single centre has been designed. Sample size will be 25.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* if woman, no pregnancy ongoing
* muscular lesion grade 2 or 3 in a lower limb muscular group

Exclusion Criteria:

* no hematological conditions
* no anticoagulation in the two preceding weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
number (and proportion with 95% CI) of patients able to return to sport activity (i.e. training) at 21 days from muscular injury. | 21 days from enrollment
  If the athlete is able, 21 days after the muscular injury, to return to (at least) training activities, the outcome will be coded "successful"; and "unsuccessful" otherwise

SECONDARY OUTCOMES:
Time-to-return to sport activities | within 4 months from lesion
Side effects | within 4 months from treatment
  Overall frequency of patients with any adverse events (number, proportion and 95%CI)
time-to-healing at ultrasound | within 4 months from treatment
side effects | within 4 months from treatment
  types of side effects (number, proportion and 95%CI for each type of adverse events)
side effects | within 4 months from treatment
  grade of side effects (number, proportion and 95%CI for each grade of adverse events)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Ortopedica Fondazione IRCCS Policlinico San Matteo, Pavia, Italy